CLINICAL TRIAL: NCT01261442
Title: Can Ultrasound Detect Diabetic Peripheral Neuropathy?
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0435-BE
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2010-06

CONDITIONS: Distal Symmetric Polyneuropathy (DSPN)
Keywords: distal symmetric polyneuropathy; diabetic peripheral neuropathy; posterior tibial nerve; regional anesthesia; nerve conduction study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic patients with DSPN
  Interventions: Procedure: Nerve Conduction Study (NCS)
- Diabetic patients without DSPN
  Interventions: Procedure: Nerve Conduction Study (NCS)

INTERVENTIONS:
Procedure: Nerve Conduction Study (NCS) — An NCS will be performed on each patient to confirm or exclude DSPN. Following this, a systematic ultrasound examination of the posterior tibial nerve will be performed for all the patients.

SUMMARY:
The cross sectional area of posterior tibial nerve (PTN) is increased in diabetic patients with distal symmetric polyneuropathy (DSPN) as compared to diabetic patients without DSPN. This study aims to evaluate whether the cross sectional area of the Posterior Tibial Nerve (PTN) as measured by ultrasound is increased in patients with distal symmetric polyneuropathy (DSPN) as compared to diabetic patients without DSPN.

DETAILED DESCRIPTION:
Regional anesthesia is associated with a low frequency of neurologic injury that can result in permanent deficit. It is believed that patients with neuropathies might be at higher risk of injury but detailed investigation of the diabetic patient is lacking yet anesthetic practices may be altered nevertheless. This study intends to investigate the appearance and sonographic qualities, as well as electrophysiologic measures, of the posterior tibial nerve (PTN) in diabetic patients undergoing nerve conduction studies in order to compare PTN characteristics between diabetic patients with peripheral neuropathy to those without. Ultimately, we hope that ultrasound, a commonly used non-invasive tool, will be able to assist in the identification of patients at higher risk of injury from regional anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Type I diabetic patients (diagnosed more than 5 years), and type II diabetic patients scheduled for routine NCS.

Exclusion Criteria:

* Non-diabetic neuropathy caused by genetic, metabolic and inflammatory diseases as well as toxic agents and drug induced (eg. chemotherapy agents)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult diabetic patients scheduled to undergo a nerve conduction study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Association of mean cross-sectional area of the PTN, as measured by sonographic imaging, with the presence of DSPN in diabetic patients. | 30 minutes

SECONDARY OUTCOMES:
Association of mean cross-sectional area of the PTN, and the severity of DSPN (graded mild, moderate, and severe) in diabetic patients with peripheral neuropathy. | 30 minutes
Descriptive sonographic appearance of PTN (ie. focal compression, hypo/hyper echogenicity, and texture). | 30 minutes
Association of mean cross-sectional area of the PTN, and the severity of DSPN (graded mild, moderate, and severe) in diabetic patients with peripheral neuropathy. | 30 minutes
  The criteria for assessment of severity of DSPN is as follows:
  1. No neuropathy: diabetic patients with no sign or symptoms of neuropathy, and normal NCS;
  2. Incipient neuropathy: diabetic patients with signs, and symptoms of neuropathy, and normal NCS;
  3. Subclinical neuropathy: Diabetic patients without signs of symptoms of neuropathy and abnormal NCS;
  4. Moderate neuropathy: diabetic patients with signs and symptoms of neuropathy and abnormal NCS;
  5. Severe neuropathy: diabetic patients with signs and symptoms of neuropathy and abnormal NCS, with absence of the sural nerve response.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada